CLINICAL TRIAL: NCT00131196
Title: Functional Genomic Influences on Disease Progression and Outcome in Sepsis Due to Pneumonia or Peritonitis
Brief Title: Functional Genomic Influences on Disease Progression and Outcome in Sepsis
Acronym: GAinS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Sainsbury Family Charitable Trusts (Other); Wellcome Trust (Other); Queen Mary University of London (Other); Barts and the London School of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Dr CS Garrard, Consultant in Intensive care, University of Oxford
Other Study IDs: N8518
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Pneumonia; Peritonitis
Keywords: pneumonia; peritonitis; sepsis; outcome; genomics
MeSH Terms: conditions — Pneumonia; Peritonitis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma and extracted DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposal is aimed at identifying genetic factors that determine the incidence and severity of, and the outcome from life-threatening infections (severe sepsis/septic shock) in patients admitted to High Dependency Units (HDUs) or Intensive Care Units (ICUs) with pneumonia which developed outside the hospital (community acquired pneumonia - CAP) or contamination of the abdominal cavity with faeces due to a leak in the bowel (faecal peritonitis). This will require the acquisition of a large, high quality resource of genetic material (DNA), plasma, urine, white blood cells and clinical information from well characterized groups of similar patients with, or at risk for, severe sepsis/septic shock. The principal objective is to perform studies which are sufficiently large to establish beyond doubt the influence of a series of selected "candidate" genes on the development, progress and outcome of sepsis.

DETAILED DESCRIPTION:
The investigators plan to recruit 2,000 cases of community acquired pneumonia (CAP) and 2,000 cases of faecal peritonitis (FP) from 30 UK ICUs and HDUs (members of the UK Critical Care Genomics group - UKCCG). The large number of patients is required to satisfy the power calculations based upon the predicted allele frequencies of candidate genes and the level of functional expression of the gene polymorphisms.

If a patient is eligible, written, informed consent will be obtained either from the patient or, if the patient is incompetent via the patient's legal representative. Patients will be characterized clinically in terms of admission diagnosis, severity of illness (APACHE II), organ failures (SOFA) and final outcome (ICU and hospital mortality, death or survival 6 months following ICU admission. Date of death will be recorded when appropriate). Clinical status will be assessed daily for days 1, 2, 3, 5 and 7 of ICU admission using the Sepsis criteria, SOFA score, microbiological culture results and antibiotic therapy.

Selected ICUs will, following consent, also undertake blood and urine sampling on days 1, 3 and 5 for genomic, proteomic and metabolomic studies. Information will be recorded on a bar-coded paper clinical report form (CRF) at the bedside. The CRFs will be securely stored locally and copied to the research coordinator, where they will be archived. The data will be entered independently by the research coordinator and one of the investigators into a secure, central web-based electronic database for storage of clinical data and the calculation of derived values. The patient codes for genetic analysis will be derived directly from the clinical database. Those undertaking genotyping will be blinded to the clinical details and these two databases will be brought together at the time of analysis only under the direct supervision of one of the principal investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patient, or legal representative, is able to give informed consent
* Male or female of 18 years or more
* Patient admitted to ICU/HDU with faecal peritonitis or community acquired pneumonia

Exclusion Criteria:

* Patient or legal representative is unwilling to consent
* Patient is under the age of 18 years
* Patient is already enrolled in an interventional study
* Patient is immunocompromised
* Patient is pregnant
* There is an advance directive to withhold or withdraw life-sustaining treatment or patient is admitted for palliative care only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care Units or High Dependency Units in the UK with faecal peritonitis or community acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2005-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
ICU and hospital Mortality | ICU discharge, hospital discharge and 6 month. The date of death will be recorded, as appropriate, for each patient.

SECONDARY OUTCOMES:
Severity of illness, duration of organ support, shock reversal, duration of ICU and hospital stay | From ICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Garrard, MD PhD, Principal Investigator — University of Oxford, UK; Charles J Hinds, MD, Principal Investigator — Queen Mary College, University of London, UK; Simon Baudouin, MD, Principal Investigator — Royal Victoria Infirmary and Freeman Hospital, Newcastle, UK; David Higgins, MD, Principal Investigator — Southend General Hospital, Southend, UK.; Richard Venn, MD, Principal Investigator — Worthing and Southlands Hospitals NHS Trust, Worthing, UK.; David Watson, MD, Principal Investigator — Homerton University Hospital, London, UK.; Atul Kapila, MD, Principal Investigator — Royal Berkshire Hospital, Reading, UK.; Simon Fletcher, MD, Principal Investigator — Norfolk and Norwich University Hospitals, Norwich, UK.; Andrew Johnston, MD, Principal Investigator — Addenbrooke's Hospital, Cambridge, UK.; Julian Bion, Professor, Principal Investigator — Queen Elizabeth Hospital, Birmingham, UK.; Gary Mills, MD, Principal Investigator — Royal Halamshire Hospital, Sheffield, UK.; Stephen Bonner, MD, Principal Investigator — James Cook University Hospital, Middlesborough, UK.; Mark Garfield, MD, Principal Investigator — The Ipswich Hospital, Ipswich, UK.; Ronald Baillie, MD, Principal Investigator — Antrim Hospital, Antrim, Northern Ireland.; George Findlay, MD, Principal Investigator — University Hospital of Wales, Cardiff,UK.; Geoffrey Bellingan, MD, Principal Investigator — UCLH Middlesex Hospital, London, UK.; Tony Gordon, MD, Principal Investigator — Charing Cross Hospital, London, UK.; Michelle Hayes, MD, Principal Investigator — Chelsea and Westminster Hospital, London, UK.; Dilshan Arawwawala, MD, Principal Investigator — Broomfield Hospital, Chelmsford, UK.; Andrew Bentley, MD, Principal Investigator — Wythenshawe Hospital, Manchester, UK.; Gareth Thomas, MD, Principal Investigator — Hope Hospital, Manchester, UK.; Julian Knight, MD, Principal Investigator — Wellcome Trust; Jonathan Thompson, MD, Principal Investigator — University Hospitals, Leicester; Jasmeet Soar, MD, Principal Investigator — Frenchay Hospital and Southmead Hospital, Bristol; Phil Watt, MD, Principal Investigator — Kettering General Hospital; Anton Krige, MD, Principal Investigator — Royal Blackburn Hospital; Ian Smith, MD, Principal Investigator — Castle Hill Hospital and Hull Royal Infirmary; Achyut Guleri, MD, Principal Investigator — Blackpool Victoria Hospital; Shond Laha, MD, Principal Investigator — Royal Preston Hospital; Stephen Brett, MD, Principal Investigator — Hammersmith Hospitals NHS Trust; Jeronimo Moreno Cuesta, MD, Principal Investigator — North Middlesex University Hospital; Pyda Venkatesh, MD, Principal Investigator — Coventry University Hospital; Peter Hall, MD, Principal Investigator — Huddersfield Royal Infirmary and Calderdale Royal Hospital; Martin Kuper, MD, Principal Investigator — The WhittingtonHospital, London. UK; Sia Pesian, MD, Principal Investigator — Manor Hospital, Walsall. UK; Andrew Timmins, MD, Principal Investigator — Colchester Hospital, Colchester . UK; Stephen Drage, MD, Principal Investigator — Royal Sussex County Hospital; Martin Stotz, MD, Principal Investigator — St. Mary's Hospital, London, UK; Mark Blunt, MD, Principal Investigator — Queen Elizabeth Hospital, King's Lynn. UK; Nigel Webster, Professor, Principal Investigator — Aberdeen Royal Infirmary; Jane Minton, MD, Principal Investigator — St James Hospital, Leeds. UK; Matt Oram, MD, Principal Investigator — Cheltenham General Hospital, Cheltenham. UK; Ingrid Krupe, MD, Principal Investigator — Lewisham Hospital; Abhiram Mallick, MD, Principal Investigator — Leeds General Infirmary, Leeds. UK; Samuel Pambakian, MD, Principal Investigator — Frimley Park Hospital, Frimley. UK; Malcolm Watters, MD, Principal Investigator — Great Western Hospital, Swindon. UK
Locations (50):
- United Kingdom (50):
  - Southmead Hospital, Bristol, Avon
  - Royal Berkshire Hospital, Reading, Berkshire
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - James Cook University Hospital, Middlesbrough, Cleveland
  - Antrim Hospital, Antrim, County Antrim
  - Castle Hill Hospital, Cottingham, East Riding of Yorkshire
  - Broomfield Hospital, Chelmsford, Essex
  - Colchester General Hospital, Colchester, Essex
  - Southend General Hospital, Southend, Essex
  - Bristol Royal Infirmary, Bristol, Gloucestershire
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Withington Hospital, Manchester, Greater Manchester
  - Wythenshawe Hospital, Manchester, Greater Manchester
  - Hope Hospital, Manchester, Greater Manchester
  - Royal Blackburn Hospital, Blackburn, Lancashire
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Royal Preston Hospital, Preston, Lancashire
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - University Hospital Lewisham, Lewisham, London
  - Queen Elizabeth Hospital, Kings Lynn, Norfolk
  - Norfolk and Norwich University Hospitals, Norwich, Norfolk
  - Kettering General Hospital, Kettering, Northants
  - John Radcliffe Hospital, Oxford, Oxon
  - University Hospital of Wales, Cardiff, South Glamorgan
  - Frenchay Hospital, Bristol, South Gloucestershire
  - The Ipswich Hospital, Ipswich, Suffolk
  - Frimley Park Hospital, Frimley, Surrey
  - Royal Sussex County Hospital, Brighton, Sussex
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - University Hospital, Coventry, Warwickshire
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Walsall Manor Hospital, Walsall, West Midlands
  - Worthing and Southlands Hospitals NHS Trust, Worthing, West Sussex
  - Calderdale Royal Hospital, Halifax, West Yorkshire
  - Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire
  - Hull Royal Infirmary, Hull, Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Glenfield Hospital, Leicester
  - Leicester General Hospital, Leicester
  - Homerton Hospital, London
  - St Bartholomew's Hospital, London
  - North Middlesex University Hospital, London
  - Chelsea and Westminster Hospital, London
  - Hammersmith Hospital, London
  - UCLH Middlesex Hospital, London
  - St Mary's Hospital, London
  - Charing Cross Hospital, London
  - Royal Halamshire Hospital, Sheffield
  - The Great Western Hospital, Swindon

REFERENCES:
- [Background] Vincent JL, Angus D, Annane D, Bernard G, Faist E, Giroir B, Reinhart K. Clinical expert round table discussion (session 5) at the Margaux Conference on Critical Illness: outcomes of clinical trials in sepsis: lessons learned. Crit Care Med. 2001 Jul;29(7 Suppl):S136-7. doi: 10.1097/00003246-200107001-00040. No abstract available. PMID 11445749
- [Background] Brun-Buisson C, Doyon F, Carlet J, Dellamonica P, Gouin F, Lepoutre A, Mercier JC, Offenstadt G, Regnier B. Incidence, risk factors, and outcome of severe sepsis and septic shock in adults. A multicenter prospective study in intensive care units. French ICU Group for Severe Sepsis. JAMA. 1995 Sep 27;274(12):968-74. PMID 7674528
- [Background] File TM. Community-acquired pneumonia. Lancet. 2003 Dec 13;362(9400):1991-2001. doi: 10.1016/S0140-6736(03)15021-0. PMID 14683661
- [Background] Gordon AC, Lagan AL, Aganna E, Cheung L, Peters CJ, McDermott MF, Millo JL, Welsh KI, Holloway P, Hitman GA, Piper RD, Garrard CS, Hinds CJ. TNF and TNFR polymorphisms in severe sepsis and septic shock: a prospective multicentre study. Genes Immun. 2004 Dec;5(8):631-40. doi: 10.1038/sj.gene.6364136. PMID 15526005
- [Background] Mira JP, Cariou A, Grall F, Delclaux C, Losser MR, Heshmati F, Cheval C, Monchi M, Teboul JL, Riche F, Leleu G, Arbibe L, Mignon A, Delpech M, Dhainaut JF. Association of TNF2, a TNF-alpha promoter polymorphism, with septic shock susceptibility and mortality: a multicenter study. JAMA. 1999 Aug 11;282(6):561-8. doi: 10.1001/jama.282.6.561. PMID 10450718
- [Background] Sands KE, Bates DW, Lanken PN, Graman PS, Hibberd PL, Kahn KL, Parsonnet J, Panzer R, Orav EJ, Snydman DR, Black E, Schwartz JS, Moore R, Johnson BL Jr, Platt R; Academic Medical Center Consortium Sepsis Project Working Group. Epidemiology of sepsis syndrome in 8 academic medical centers. JAMA. 1997 Jul 16;278(3):234-40. PMID 9218672
- [Background] Sorensen TI, Nielsen GG, Andersen PK, Teasdale TW. Genetic and environmental influences on premature death in adult adoptees. N Engl J Med. 1988 Mar 24;318(12):727-32. doi: 10.1056/NEJM198803243181202. PMID 3347221
- [Background] Roy S, Knox K, Segal S, Griffiths D, Moore CE, Welsh KI, Smarason A, Day NP, McPheat WL, Crook DW, Hill AV; Oxford Pneumoccocal Surveillance Group. MBL genotype and risk of invasive pneumococcal disease: a case-control study. Lancet. 2002 May 4;359(9317):1569-73. doi: 10.1016/S0140-6736(02)08516-1. PMID 12047967
- [Derived] Scicluna BP, Cano-Gamez K, Burnham KL, Davenport EE, Moore AR, Khan S, Hinds CJ, Cremer OL, Khatri P, Sweeney TE, Knight JC, van der Poll T. A consensus blood transcriptomic framework for sepsis. Nat Med. 2025 Dec;31(12):4119-4130. doi: 10.1038/s41591-025-03964-5. Epub 2025 Sep 30. PMID 41028542
- See also: GAinS Website (Genomic Advances in Sepsis) — http://www.ukccg-gains.org/